CLINICAL TRIAL: NCT01977677
Title: A Phase I/II Study of Local Field Irradiation and Temozolomide Followed by Continuous Infusion Plerixafor as an Upfront Therapy for Newly Diagnosed Glioblastoma GBM
Brief Title: Plerixafor After Radiation Therapy and Temozolomide in Treating Patients With Newly Diagnosed High Grade Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Lawrence Recht (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Lawrence Recht, Professor of Neurology, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRN0023; NCI-2013-02012 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BRN0023 (Other: Stanford University Hospitals and Clinics); P30CA124435 (NIH)
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Results first posted 2018-07-03 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-09

CONDITIONS: Adult Ependymoblastoma; Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Medulloblastoma; Adult Mixed Glioma; Adult Oligodendroglial Tumors; Adult Pineoblastoma; Adult Supratentorial Primitive Neuroectodermal Tumor (PNET)
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive; Glioblastoma; Gliosarcoma; Medulloblastoma; Glioma; Pinealoma | interventions — Radiotherapy; Radiation; Temozolomide; plerixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (radiation therapy, temozolomide, plerixafor) (Experimental): Within 4 weeks of surgery, patients undergo radiation therapy and receive temozolomide PO over 42 days. Beginning 8 days prior to completion of chemoradiotherapy, patients receive plerixafor IV continuously for 2-4 weeks. Patients also receive temozolomide PO 5 days a month beginning 35 days after completion of radiation therapy.
  Interventions: Radiation: radiation therapy; Drug: temozolomide; Drug: plerixafor; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: temozolomide — Given PO
  Other Names: SCH 52365; Temodal; Temodar; TMZ
Drug: plerixafor — Given IV
  Other Names: AMD 3100; Mozobil
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This pilot phase I/II trial studies the side effects and best dose of plerixafor after radiation therapy and temozolomide and to see how well it works in treating patients with newly diagnosed high grade glioma. Plerixafor may stop the growth of tumor cells by blocking blood flow to the tumor. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high energy x rays to kill tumor cells. Giving plerixafor after radiation therapy and temozolomide may be an effective treatment for high grade glioma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of using continuous infusion Plerixafor subsequent to irradiation in patients with newly diagnosed glioblastoma multiforme (GBM).

II. To assess the efficacy of Plerixafor as measured by progression free survival at 6 months (PFS6) from the start of irradiation.

OUTLINE: This is a phase I, dose-escalation study of plerixafor followed by a phase II study.

Within 4 weeks of surgery, patients undergo radiation therapy and receive temozolomide orally (PO) over 42 days. Beginning 8 days prior to completion of chemoradiotherapy, patients receive plerixafor intravenously (IV) continuously for 2-4 weeks. Patients also receive temozolomide PO 5 days a month beginning 35 days after completion of radiation therapy.

After completion of study treatment, patients are followed up every 12 weeks for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have tissue confirmation of high grade (WHO Grade IV) glioma including but not limited to glioblastoma, gliosarcoma, glioblastoma with oligodendroglial features, glioblastoma with PNET features.
* The patient must have post-operative contrast enhanced imaging (CT or MRI) unless only biopsy performed (in which case post-operative imaging is not routinely obtained. In these patients, the preoperative study will serve as baseline.
* Patient should have surgery (biopsy, partial resection or gross total resection) and no additional anti-cancer therapy except the chemoradiation as specified in the protocol.
* For those patients in which steroids are clinically indicated, there must be a stable or decreasing dose of steroid medication for ≥ one week prior to the start of infusion.
* Patients must be between the ages of 18 and 75 years old.
* Patients must have Karnofsky Performance score ≥ 60.
* Adequate organ function is needed at time of screening visit including:

  * ANC ≥ 1500
  * Platelets ≥ 100,000 ml
  * Serum Creatinine ≤ 1.5mg/dl; Cr Clearance should be >50 mL/min
  * AST and ALT ≤ 3 times the upper limit of normal
  * If female of childbearing potential, negative pregnancy test
* The patient or his/her legal representative must have the ability to understand and willingness to sign a written informed consent document.
* Patient agrees to use an effective method of contraception (hormonal or two barrier methods) while on study and for at least 3 months following the Plerixafor infusion

Exclusion Criteria:

* Prior or concurrent treatment with Avastin (bevacizumab)
* Prior exposure to Plerixafor
* Prior use of other investigational agents to treat the brain tumor
* Recent history of myocardial infarct (less than 3 months) or history of active angina or arrhythmia
* Prior malignancy except previously diagnosed and definitively treated more than 3 years prior to trial or whose prognosis is deemed good enough to not warrant surveillance
* Prior sensitivity to Plerixafor
* Pregnant or patients who are breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-11; Primary Completion 2017-11 (Actual); Study Completion 2018-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Recht, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 30 patients were enrolled at one study center.
Pre-assignment Details: A total of 32 subjects were screened. One was a screen failure, one withdrew consent prior to initiating the infusion. Twenty-nine subjects enrolled and completed the 28 day Plerixafor infusion. One subject enrolled but did not complete the infusion due to an unrelated adverse event.
Groups:
- Escalation: Plerixafor 200 mcg/kg/Day: One week prior to the completion of radiotherapy with concurrent temozolomide, patients with newly diagnosed glioblastoma will receive continuous infusion of Plerixafor at a dose of 200 mcg/kg/day over 4 weeks.
- Escalation: Plerixafor 400 mcg/kg/Day; Expansion: Plerixafor 400 mcg/kg/Day: One week prior to the completion of radiotherapy with concurrent temozolomide, patients with newly diagnosed glioblastoma will receive continuous infusion of Plerixafor at a dose of 400 mcg/kg/day over 4 weeks.
Period: Overall Study
Arm/Group | Escalation: Plerixafor 200 mcg/kg/Day | Escalation: Plerixafor 400 mcg/kg/Day | Expansion: Plerixafor 400 mcg/kg/Day
Started | 3 | 6 | 21
Completed | 3 | 6 | 20
Not Completed | 0 | 0 | 1
Not completed — Unrelated Adverse Event | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Only subjects who completed the 4 week infusion were included
Groups:
- Total: Total of all reporting groups
Arm/Group | Escalation: Plerixafor 200 mcg/kg/Day | Escalation: Plerixafor 400 mcg/kg/Day | Expansion: Plerixafor 400 mcg/kg/Day | Total
Number analyzed (Participants) | 3 | 6 | 20 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 15 | 20
  >=65 years | 1 | 3 | 5 | 9
Age, Continuous [Median (Full Range); unit: years] | 64 [55 to 67] | 62 [40 to 74] | 60 [29 to 74] | 60 [29 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 9
  Male | 1 | 4 | 15 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 6 | 19 | 28
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 4 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 3 | 5 | 14 | 22
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 20 | 29

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicity
Description: Dose Limiting Toxicity is defined as defined as any hematologic or on-hematologic adverse events grade 3 or higher using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 with a suspected causal relationship to Plerixafor (including electrocardiogram changes indicative of ischemia, ventricular tachycardia)
Time Frame: Up to 30 days post plerixafor
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation: Plerixafor 200 mcg/kg/Day | Escalation: Plerixafor 400 mcg/kg/Day | Expansion: Plerixafor 400 mcg/kg/Day
Number analyzed (Participants) | 3 | 6 | 21
Participants | 0 | 0 | 0

2. Primary Outcome: Participants Alive and Without Disease Progression At 6 Months After the Start of the Irradiation
Description: Progression free survival based on the Response Assessment for Neuro-Oncology (RANO) criteria, using both clinical examinations and MRIs with and without contrast summarized with Kaplan Meier estimates.
Time Frame: 6 months from start of irradiation
Measure: Count of Participants; unit: Participants
Arm/Group | Escalation: Plerixafor 200 mcg/kg/Day | Escalation: Plerixafor 400 mcg/kg/Day | Expansion: Plerixafor 400 mcg/kg/Day
Number analyzed (Participants) | 3 | 6 | 20
Participants | 3 | 5 | 19

ADVERSE EVENTS:
Time Frame: Up to 30 days after Plerixafor Infusion
Arm/Group | Escalation: Plerixafor 200 mcg/kg/Day | Escalation: Plerixafor 400 mcg/kg/Day | Expansion: Plerixafor 400 mcg/kg/Day
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/6 | 1/21
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/6 | 3/21
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6 | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escalation: Plerixafor 200 mcg/kg/Day (N=3) | Escalation: Plerixafor 400 mcg/kg/Day (N=6) | Expansion: Plerixafor 400 mcg/kg/Day (N=21)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Disease Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Pseudoprogression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Hemorrhagic hepatic cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escalation: Plerixafor 200 mcg/kg/Day (N=3) | Escalation: Plerixafor 400 mcg/kg/Day (N=6) | Expansion: Plerixafor 400 mcg/kg/Day (N=21)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral dysesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 4 (4)
Parasthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Cognitive Disturbance (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Facial Muscle Weakness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Memory Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 4 (4) | 7 (7)
Confusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucinations (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Bad dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 1 (1) | 6 (6)
Gait Disturbance (General disorders) | 0 (0) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Localized Edema (General disorders) | 0 (0) | 0 (0) | 1 (1)
Hot Flashes (Vascular disorders) | 1 (1) | 2 (2) | 5 (5)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Cardiac Troponin 1 increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
INR increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
White blood cell decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
wart like growth (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Bullous Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 3 (3) | 0 (0)
Dry Eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye Pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Watering Eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Bone infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Thrush (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Allergic Reaction (Immune system disorders) | 1 (1) | 1 (1) | 0 (0)
Enhanced immune response (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Allergic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash Spots on head (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT01977677/Prot_SAP_000.pdf